CLINICAL TRIAL: NCT04505618
Title: Optical Coherence Tomography Angiography in Subjects With Retinal Vascular Disease
Acronym: OCTA-RVD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB00276904; R01EY030564 (NIH)
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2025-06-16 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Retinopathy; Retinal Vein Occlusion; Hypertension,Essential; Retinal Vascular Disorder
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Vein Occlusion; Essential Hypertension | interventions — Optical Imaging; Lenses, Intraocular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Controls (Other): Subjects in this group do not have any ocular pathology and are also not hypertensive. Some subjects in this arm will undergo retinal vascular reactivity assessments.
  Interventions: Device: Swept-Source (SS) OCT Angiography; Device: Spectral-Domain (SD) OCT Angiography; Device: Fundus Imaging; Device: Axial Length Measurement Device
- Diabetics with and without Diabetic Retinopathy Only (Other): Subjects in this group only have diabetes with or without diabetic retinopathy. Some subjects in this arm will undergo retinal vascular reactivity assessments.
  Interventions: Device: Swept-Source (SS) OCT Angiography; Device: Spectral-Domain (SD) OCT Angiography; Device: Fundus Imaging; Device: Axial Length Measurement Device
- Hypertension Only (Other): Subjects in this group only have hypertension with or without ocular pathology related to hypertension. Some subjects in this arm may undergo retinal vascular reactivity assessments.
  Interventions: Device: Swept-Source (SS) OCT Angiography; Device: Spectral-Domain (SD) OCT Angiography; Device: Fundus Imaging; Device: Axial Length Measurement Device
- Diabetics w/ or w/o Diabetic Retinopathy & Hypertension (Other): Subjects in this group have diabetes with or without diabetic retinopathy and hypertension with or without ocular pathology related to hypertension. Some subjects in this arm may undergo retinal vascular reactivity assessments.
  Interventions: Device: Swept-Source (SS) OCT Angiography; Device: Spectral-Domain (SD) OCT Angiography; Device: Fundus Imaging; Device: Axial Length Measurement Device

INTERVENTIONS:
Device: Swept-Source (SS) OCT Angiography — Non-invasive, minimal risk, ocular imaging study
  Other Names: SS-OCTA
Device: Spectral-Domain (SD) OCT Angiography — Non-invasive, minimal risk, ocular imaging study
  Other Names: SD_OCTA
Device: Fundus Imaging — Non-invasive, minimal risk, ocular imaging study
Device: Axial Length Measurement Device — Non-invasive, minimal risk, ocular imaging study
  Other Names: Intraocular Lens (IOL) Master

SUMMARY:
This study will perform a prospective, longitudinal analysis of clinical and imaging findings from normal controls and subjects with retinal vascular disease to better define the diagnostic imaging criteria that signify change in disease stage. This includes disease progression in early stages of disease or disease regression with appropriate standard-of-care treatment.

DETAILED DESCRIPTION:
The objective of this study is to perform a prospective, longitudinal analysis of clinical and imaging findings from normal controls and subjects with retinal vascular disease to better define the diagnostic imaging criteria that signify change in disease stage. This includes disease progression in early stages of disease or disease regression with appropriate standard-of-care treatment.

Subjects will be identified from healthy subjects (seen for screening eye exams) and diseased subjects undergoing standard-of-care treatment or screening at eye clinic locations. The study population will include subjects with retinal vascular disease including but not limited to diabetic retinopathy, hypertension, retinal vein/arterial occlusion, and macular degeneration. Subjects who are enrolled will undergo non-invasive, minimal risk, FDA approved diagnostic imaging procedures to identify vascular changes.

The study methods will include retrospective review and collection of clinically approved imaging data that is obtained through standard-of-care methods for subjects who meet inclusion and exclusion criteria. Subjects who are identified in this manner will be asked to participate in a prospective study by each clinical study site.

The study end-points include the correlation of diagnostic imaging findings from Optical Coherence Tomography (OCT) based images with fundus photographs, clinical disease stage and visual acuity.

ELIGIBILITY:
Exclusion Criteria:

* Both subjects with diseases and controls:
* Children (age<18)
* Pregnant females
* Developmentally delayed subjects
* Subjects unable to provide informed consent
* Inability to cooperate with tests and study instructions
* Images with motion artifact or signal strength < 7
* History of glaucoma
* History of age-related macular degeneration
* History of any visually significant eye disease
* History of proliferative diabetic retinopathy
* History of any inflammatory disease
* History of heart disease
* History of thyroid disease.
* Additional criteria for controls:
* History of any type of Diabetes Mellitus
* History of any type of Hypertension

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of Imaging | 5 years
  Correlation of diagnostic imaging findings (vessel skeleton density) from OCT based images with disease stage

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kashani, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States